CLINICAL TRIAL: NCT00616655
Title: A Double Blind, Randomized, Placebo Controlled, Multicenter Study Examining the Efficacy and Safety of SEP-225441 in Subjects With Generalized Anxiety Disorder.
Brief Title: Generalized Anxiety Disorder Proof of Concept Efficacy and Safety Study of SEP-225441 (Eszopiclone) In GAD Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 194-027
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): SEP-225441 (eszopiclone) total daily dose of 1.5 mg
  Interventions: Drug: eszopiclone
- 2 (Active Comparator): SEP-225441 (eszopiclone) total daily dose of 0.9 mg
  Interventions: Drug: eszopiclone
- 3 (Placebo Comparator): Placebo total daily dose 0.9 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eszopiclone — SEP-225441 (eszopiclone) total daily dose of 1.5 mg
  Other Names: SEP-225441
  Arms: 1
Drug: eszopiclone — SEP-225441 (eszopiclone) total daily dose of 0.9 mg
  Other Names: SEP-225441
  Arms: 2
Drug: Placebo — Placebo total daily dose 0.9 mg
  Arms: 3

SUMMARY:
To determine the safety and efficacy of SEP-225441 (eszopiclone) in subjects with generalized anxiety disorder (GAD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double blind, placebo controlled study of the safety and efficacy of SEP-225441 (eszopiclone) in male and female adult subjects with a diagnosis of generalized anxiety disorder (GAD). The study consists of a screening period of 7-10 days, 8 weeks of treatment, and a 7 day follow-up period. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be between 18 and 50 years of age
* Subjects must have GAD
* Subjects must be in otherwise good general health

Exclusion Criteria:

* Subject has a documented history of HIV, hepatitis B or hepatitis C.
* Subject has a recent history (within 6 months of study entry) or current diagnosis of Major Depressive Disorder, panic disorder (or 3 or more panic attacks in the past month). Post Traumatic Stress Disorder, body dysmorphic disorder, eating disorder, or other disorder.
* Subject has a history or presence of Obsessive-Compulsive Disorder (OCD), any psychotic, bipolar or schizophrenic disorder.
* Subject has presence or history of antisocial personality or other severe disorder
* Subject has refractory GAD (previously unresponsive to 2 or more adequate courses of SSRI, SNRI, benzodiazepine or non-benzodiazepine treatment for GAD).
* Subject has history of seizures, including febrile seizures.
* Subject has initiated psychotherapeutic intervention with 30 days; however, continued psychotherapy is allowed if stable and not specifically directed at GAD.
* Subject is undergoing or has undergone electroconvulsive therapy.
* Subject is a current smoker or has smoked within the last 12 months.
* Subject has donated blood within the past 30 days or plans to donate during and within 30 days after study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 456 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (57):
- United States (57):
  - Birmingham Psychiatry Pharaceutical Studies, Inc., Birmingham, Alabama
  - Arcadia, California
  - Southwestern Research, Inc., Beverly Hills, California
  - Southwestern Research, Inc., Burbank, California
  - California Clinical Trials Medical Group, Glendale, California
  - California clinical Trials Medical Group, Glendale, California
  - Newport Beach, California
  - Excell Research, Oceanside, California
  - California Clinical Trials Medical Group, Paramount, California
  - Southwestern Research, Inc., Pasadena, California
  - California clinical Trials Medical Group, San Diego, California
  - Stanford Universtiy Medical center, Stanford, California
  - University of CT Health Center, Farmington, Connecticut
  - Comprehensive Psychiatric Care, PC, Norwich, Connecticut
  - Florida Clinical Research Center LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainsville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Comprehensive NeuroScience, Inc., Atlanta, Georgia
  - Carmen Research, Smyrna, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Comprehensive NeuroScience, Inc., Park Ridge, Illinois
  - Vince and Associats Clinical Research, Overland Park, Kansas
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Pedia Research, LLC, Owensboro, Kentucky
  - Pharasite Research, Inc., Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Coastal Research Associates, Inc., Braintree, Massachusetts
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - CRI Worldwide, LLC, Clementon, New Jersey
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Comprehensive NeuroScience, Inc., Fresh Meadows, New York
  - Fieve Clinica Services, Inc., New York, New York
  - Medical & Behavioral Health Research, PC, New York, New York
  - Medical & Behavioral Health Research, P.C., New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Glenwood Psychiatric Associates, P.L.L.C., Raleigh, North Carolina
  - Horizon Medical Services, Bismarck, North Dakota
  - North Coast Clinical Trials, Beachwood, Ohio
  - Patient Priority Clinical Sties, LLC, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - North Star Mdical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Eugene, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Future Search Trials, Austin, Texas
  - Carolos Guerra, Jr., M.D., Houston, Texas
  - San Antonio Psychiatric Research Center, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - University of Virginia, Center for Psychiatric Clinical Research, Charlottesville, Virginia

REFERENCES:
- [Derived] Williams JB, Kobak KA, Giller E, Reasner DS, Curry L, Detke MJ. Comparison of Site-Based Versus Central Ratings in a Study of Generalized Anxiety Disorder. J Clin Psychopharmacol. 2015 Dec;35(6):654-60. doi: 10.1097/JCP.0000000000000422. PMID 26488677

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Arm: Placebo
- Eszopiclone Low Dose Arm: SEP-225441 (eszopiclone) total daily dose of 0.9 mg
- Eszopiclone High Dose Arm: SEP-225441 (eszopiclone) total daily dose of 1.5 mg
Period: Overall Study
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Started | 152 | 153 | 151
Completed | 117 | 112 | 103
Not Completed | 35 | 41 | 48
Not completed — Adverse Event | 10 | 7 | 12
Not completed — Lack of Efficacy | 5 | 5 | 5
Not completed — Lost to Follow-up | 3 | 12 | 10
Not completed — Protocol Violation | 2 | 4 | 3
Not completed — Withdrawal by Subject | 9 | 7 | 11
Not completed — Does not meet in/ex criteria | 0 | 0 | 2
Not completed — Other | 6 | 6 | 5

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm | Total
Number analyzed (Participants) | 149 | 146 | 145 | 440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 149 | 146 | 145 | 440
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 108 | 102 | 321
  Male | 38 | 38 | 43 | 119
Region of Enrollment [Number; unit: participants]
  United States | 149 | 146 | 145 | 440

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the Total Score on the Hamilton Anxiety Scale (HAM-A), as Assessed by the Site-trained Rater
Description: THe HAM-M was administered by a site-trained rater and measured the severity of the subjects' anxiety symptoms using 14 items of the HAM-M rating scale. These items included: anxious mood, tension, fears, insomnia, intellectual, depressed mood, somatic complaints-muscular, somatic complaints-sensory, cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms, and behavior at interview. All items are measured on a 5-point scale (0-4). The Ham-A total score can range from 0 to 56 with higher scores indicating higher severity of anxiety symptoms.
Time Frame: Baseline to Week 8
Population: ITT Population: /The ITT population will include all randomized subjects who received at least one does of study medication during the double-blind period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
Units on a scale | -10.0 (7.0) | -9.3 (7.4) | -9.5 (8.1)

2. Secondary Outcome: Change From Baseline Hamilton Anxiety Scale (HAM-A) Total Score (Except for Week 8)
Description: The HAM-A was administered by a site-trained rater and measured the severity of the subjects' anxiety symptoms using 14 items of the HAM-A rating scale. These items included: anxious mood, tension, fears, insomnia, intellectual, depressed mood, somatic complaints-muscular, somatic complaints-sensory, cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms, and behavior at interview. all items are measured on a 5-point scale (0-4). Ham-A total score can range from 0 to 56 with higher scores indicating higher severity of anxiety symptoms.
Time Frame: Baseline, Weeks 2, 4, 6 based on last observation carried forward (LOCF)
Population: ITT Population: The ITT population will include all randomized subjects who received at least one dose of study medication during the double-blind period.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
unit on a scale
  Baseline | 24.2 (3.4) | 24.0 (3.4) | 24.0 (3.7)
  Week 2 - Change from baseline | -5.7 (5.7) | -4.8 (5.0) | -6.0 (6.1)
  Week 4-Change from baseline | -8.1 (6.0) | -7.6 (6.3) | -8.0 (6.8)
  Week 6- Change from baseline | -8.9 (6.3) | -8.7 (7.2) | -8.5 (7.4)

3. Secondary Outcome: Change in Individual Item Scores on HAM-A
Description: The HAM-A was administered by a site trained rater and measured the severity of the subjects' anxiety symptoms using 14 items of the HAM-A rating scale. These items include: anxious mood, tension, fears, insomnia, intellectual, depressed mood, somatic complaints-muscular, somatic complaints-sensory, cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms, and behavior at interview. All items are measured on a t5-point scale (0-4). Each HAM-A individual item score can range from 0 to 4 with higher scores indicating higher severity of anxiety questions.
Time Frame: Baseline, Weeks 2, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
units on a scale
  Anxious Mood-Baseline | 2.8 (0.5) | 2.8 (0.5) | 2.8 (0.5)
  Anxious Mood-Week 2 -Change from baseline | -0.6 (0.8) | -0.5 (0.7) | -0.6 (0.9)
  Anxious Mood-Week 4 - Change from baseline | -0.8 (0.9) | -0.8 (0.8) | -0.9 (1.0)
  Anxious Mood-Week 6 - Change from baseline | -1.0 (0.9) | -0.8 (0.8) | -1.0 (1.0)
  Anxious Mood-Week 8- Change from baseline | -1.0 (1.0) | -0.9 (0.9) | -1.1 (1.1)
  Tension - Baseline | 2.7 (0.5) | 2.6 (0.5) | 2.7 (0.5)
  Tension - Week 2 -Change from baseline | -0.5 (0.9) | -0.4 (0.7) | -0.6 (0.9)
  Tension - Week 4 - Change from baseline | -0.8 (1.0) | -0.6 (0.9) | -0.8 (0.9)
  Tension - Week 6- Change from baseline | -0.9 (1.0) | -0.8 (1.0) | -1.0 (1.0)
  Tension - Week 8- Change from baseline | -0.9 (1.0) | -0.9 (1.0) | -1.0 (1.0)
  Fears- Baseline | 1.1 (1.1) | 1.2 (1.0) | 1.0 (0.9)
  Fears- Week 2- Change from baseline | -0.3 (0.9) | -0.4 (0.8) | -0.2 (0.8)
  Fears- Week 4- Change from baseline | -0.4 (0.9) | -0.5 (0.9) | -0.3 (0.8)
  Fears- Week 6- Change from baseline | -0.4 (1.0) | -0.5 (0.9) | -0.4 (0.9)
  Fears- Week 8- Change from baseline | -0.5 (0.9) | -0.7 (1.0) | -0.4 (0.9)
  Insomnia- Baseline | 2.5 (0.7) | 2.5 (0.7) | 2.6 (0.8)
  Insomnia- Week 2- Change from baseline | -0.5 (0.9) | -0.5 (1.0) | -0.8 (1.0)
  Insomnia- Week 4- Change from baseline | -0.8 (1.1) | -0.8 (1.0) | -0.9 (1.0)
  Insomnia- Week 6- Change from baseline | -0.8 (1.0) | -0.8 (1.0) | -0.9 (1.1)
  insomnia- Week 8- Change from baseline | -0.9 (1.1) | -0.8 (1.0) | -1.0 (1.2)
  Intellectual- Baseline | 2.1 (0.8) | 2.1 (0.8) | 2.2 (0.8)
  Intellectual- Week 2- Change from baseline | -0.4 (0.9) | -0.4 (0.9) | -0.5 (0.9)
  Intellectual- Week 4- Change from baseline | -0.8 (1.0) | -0.6 (0.9) | -0.7 (0.9)
  Intellectual- Week 6- Change from baseline | -0.7 (1.1) | -0.7 (1.0) | -0.8 (1.1)
  Intellectual- Week 8- Change from baseline | -0.9 (1.1) | -0.8 (1.1) | -0.9 (1.1)
  Depressed Mood- Baseline | 1.1 (0.8) | 1.2 (0.7) | 1.0 (0.7)
  Depressed Mood- Week 2- Change from baseline | -0.3 (0.8) | -0.2 (0.8) | -0.2 (0.8)
  Depressed Mood- Week 4- Change in baseline | -0.4 (0.9) | -0.3 (0.9) | -0.3 (0.8)
  Depressed Mood- Week 6- Change from baseline | -0.3 (0.9) | -0.3 (0.9) | -0.3 (0.8)
  Depressed Mood- Week 8- Change from baseline | -0.4 (0.9) | -0.4 (0.9) | -0.3 (0.9)
  Somatic Complaints-Muscular-Baseline | 2.0 (0.8) | 1.9 (0.8) | 1.8 (0.8)
  Somatic Complaints-Muscular-Wk 2-Chg from baseline | -0.5 (1.0) | -0.3 (0.8) | -0.5 (0.8)
  Somatic Complaints-Muscular-Wk 4-Chg from baseline | -0.7 (0.9) | -0.5 (1.0) | -0.6 (0.9)
  Somatic Complaints-Muscular-Wk 6-Chg from baseline | -0.8 (1.1) | -0.7 (1.1) | -0.6 (1.0)
  Somatic Complaints-Muscular-Wk 8-Chg from baseline | -0.9 (1.1) | -0.7 (1.1) | -0.7 (1.1)
  Somatic Complaints-Sensory-Baseline | 1.0 (0.9) | 1.0 (0.9) | 1.2 (0.9)
  Somatic Complaints-Sensory-Wk 2-Chg from baseline | -0.3 (0.9) | -0.2 (0.8) | -0.5 (1.0)
  Somatic Complaints-Sensory-Wk 4-Chg from baseline | -0.4 (0.9) | -0.3 (1.0) | 1.0 (0.9)
  Somatic Complaints-Sensory-Wk 6-Chg from baseline | -0.4 (0.9) | -0.4 (0.9) | -0.5 (1.0)
  Somatic Complaints-Sensory-Wk 8-Chg from baseline | -0.5 (1.0) | -0.4 (1.0) | -0.5 (1.0)
  Cardiovascular symptoms-baseline | 1.1 (1.0) | 1.2 (1.0) | 1.3 (1.0)
  Cardiovascular symptoms-Wk 2-Chg. from baseline | -0.4 (1.0) | -0.4 (0.9) | -0.5 (1.0)
  Cardiovascular symptoms-Wk 4-Chg. from baseline | -0.5 (1.0) | -0.7 (1.0) | -0.6 (1.0)
  Cardiovascular symptoms-Wk 6-Chg. from baseline | -0.6 (1.0) | -0.6 (1.0) | -0.6 (1.0)
  Cardiovascular symptoms-Wk 8-Chg. from baseline | -0.7 (1.0) | -0.8 (1.0) | -0.7 (1.1)
  Respiratory Symptoms-Baseline | 1.2 (0.9) | 1.2 (0.9) | 1.3 (0.9)
  Respiratory Symptoms-Wk 2 Change from baseline | -0.4 (0.9) | -0.3 (0.8) | -0.4 (0.9)
  Respiratory Symptoms-Wk 4 Change from baseline | -0.5 (0.9) | -0.5 (0.9) | -0.5 (1.0)
  Respiratory Symptoms-Wk 6 Change from baseline | -0.6 (0.9) | -0.5 (1.0) | -0.5 (1.1)
  Respiratory Symptoms-Wk 8 Change from baseline | -0.6 (0.9) | -0.6 (0.9) | -0.7 (1.0)
  Gastrointestinal Symptoms- Baseline | 1.4 (1.0) | 1.4 (1.0) | 1.3 (0.9)
  Gastrointestinal Symptoms-Wk2-Change from baseline | -0.3 (1.1) | -0.4 (1.0) | -0.3 (1.1)
  Gastrointestinal Symptoms-Wk4-Change from baseline | -0.5 (1.0) | -0.5 (1.0) | -0.4 (1.1)
  Gastrointestinal Symptoms-Wk6-Change from baseline | -0.6 (1.0) | -0.6 (1.0) | -0.5 (1.1)
  Gastrointestinal Symptoms-Wk8-Change from baseline | -0.6 (1.0) | -0.6 (1.0) | -0.5 (1.1)
  Genitourinary Symptoms-Baseline | 1.5 (1.0) | 1.4 (1.0) | 1.4 (1.1)
  Genitourinary Symptoms-Wk 2-Change from baseline | -0.4 (1.0) | -0.2 (1.0) | -0.3 (1.0)
  Genitourinary Symptoms-Wk 4-Change from baseline | -0.4 (1.1) | -0.4 (1.1) | -0.4 (1.1)
  Genitourinary Symptoms-Wk 6-Change from baseline | -0.5 (1.1) | -0.4 (1.1) | -0.3 (1.0)
  Genitourinary Symptoms-Wk 8-Change from baseline | -0.6 (1.1) | -0.5 (1.1) | -0.4 (1.1)
  Autonomic Symptoms-Baseline | 1.8 (0.9) | 1.8 (0.8) | 1.8 (0.8)
  Autonomic Symptoms-Wk 2-Change from baseline | -0.4 (0.9) | -0.3 (0.9) | -0.4 (1.0)
  Autonomic Symptoms-Wk 4-Change from baseline | -0.5 (1.0) | -0.5 (1.2) | -0.5 (0.9)
  Autonomic Symptoms-Wk 6-Change from baseline | -0.6 (1.0) | -0.6 (1.1) | -0.6 (1.0)
  Autonomic Symptoms-Wk 8-Change from baseline | -0.8 (1.1) | -0.7 (1.2) | -0.6 (1.0)
  Behavior at Interview-Baseline | 1.8 (0.7) | 1.8 (0.6) | 1.8 (0.6)
  Behavior at Interview-Wk 2- Change from baseline | -0.4 (0.8) | -0.3 (0.7) | -0.4 (0.8)
  Behavior at Interview-Wk 4- Change from baseline | -0.6 (0.7) | -0.6 (0.8) | -0.5 (0.7)
  Behavior at Interview-Wk 6- Change from baseline | -0.7 (0.8) | -0.7 (0.8) | -0.7 (0.8)
  Behavior at Interview-Wk 8- Change from baseline | -0.8 (0.8) | -0.6 (0.9) | -0.7 (0.9)

4. Secondary Outcome: Change From Baseline in Clinician Global Impression of Severity (CGI-S)
Description: The CGI-Swas completed by a board certified psychiatrist and represents the clinician's subjective assessment of severity of the subject's anxiety symptoms as assessed by a 7-scale score for a single question, "Considering your total clinical experience with this particular population, how anxious is the subject at this time?" The score was based on the following scale: 1=normal, not at all anxious; 2=borderline anxious; 3=mildly anxious; 4=moderately anxious; 5=markedly anxious; 6=severly anxious; 7=among the most extremely anxious subjects. CGI-S score can range from 0 to 7, with higher values indicating higher severity.
Time Frame: Baseline, Weeks 2, 4, 6, 8, based on last observation carried forward (LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
units on a scale
  Baseline | 4.4 (0.5) | 4.3 (0.5) | 4.4 (0.6)
  Week 2 - Change from baseline | -0.6 (0.9) | -0.4 (0.6) | -0.7 (0.9)
  Week 4- Change from baseline | -0.9 (0.9) | -0.8 (0.8) | -1.0 (1.1)
  Week 6- Change from baseline | -1.1 (1.0) | -1.0 (1.0) | -1.2 (1.2)
  Week 8- Change from baseline | -1.3 (1.1) | -1.2 (1.1) | -1.3 (1.3)

5. Secondary Outcome: Clinical Global Impression- Improvement (CGI-I)
Description: CGI-I was completed by a board certified psychiatrist and represented the clinician's subjective assessment of improvement of the subject's anxiety symptoms based on the following question, "Compared to his/her condition at Visit 2, how much has he/she changed?" The score was based on the following scale: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. CGI-I score can range from 0 to 7, with higher values indicating less improvement.
Time Frame: Weeks 2, 4, 6, 8, and 9, based on last observation carried forward (LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
units on a scale
  Week 2 | 3.2 (1.0) | 3.2 (0.9) | 3.1 (1.0)
  Week 4 | 2.9 (1.0) | 2.9 (0.9) | 2.7 (1.2)
  Week 6 | 2.7 (1.0) | 2.6 (1.1) | 2.7 (1.2)
  Week 8 | 2.6 (1.1) | 2.6 (1.1) | 2.6 (1.2)
  Week 9 | 2.4 (1.1) | 2.5 (1.1) | 2.4 (1.2)

6. Secondary Outcome: Hamilton Anxiety Scale (HAM-A) 50% Anxiolytic Response
Description: The HAM-A was administered by a site-trained rater and measured the severity of the subjects' anxiety symptoms using 14 items of the HAM-A rating scale. These items include: anxious mood, tension, fears, insomnia, intellectual, depressed mood, somatic complaints-muscular, somatic complaints-sensory, cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms, and behavior at interview. All items are measured on a 5-point scale (0-4). A 50% anxiolytic response was defined as a 50% or greater reduction from baseline in the HAM-A total score.
  The Ham-A total score can range from 0 to 56 with higher scores indicating higher severity of anxiety symptoms.
Time Frame: Week 2, 4, 6, 8
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
participants
  Week 2 | 21 | 16 | 27
  Week 4 | 39 | 41 | 49
  Week 6 | 51 | 52 | 53
  Week 8 | 63 | 57 | 66

7. Secondary Outcome: Hamilton Anxiety Scale (HAM-A) Remission
Description: The HAM-A was administered by a site-trained rater and measured the severity of the subjects' anxiety symptoms using 14 items of the HAM-A rating scale. These items include: anxious mood, tension, fears, insomnia, intellectual, depressed mood, somatic complaints-muscular, somatic complaints-sensory, cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms, autonomic symptoms, and behavior at interview. All items are measured on a 5-point scale (0-4). Remission was defined as a HAM-A total score of 7 or less.
  The Ham-A total score can range from 0 to 56 with higher scores indicating higher severity of anxiety symptoms.
Time Frame: Week 2, 4, 6, 8 based on last observation carried forward (LOCF)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
participants
  Week 2 | 7 | 2 | 9
  Week 4 | 11 | 10 | 24
  Week 6 | 22 | 19 | 23
  Week 8 | 31 | 29 | 34

8. Secondary Outcome: Change From Baseline on Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Short Form
Description: The Q-LES-Q was completed by the subject and assessed quaility of life based on 16 items, each evaluated on a 5-point scale of overall level of enjoyment/satisfaction: 1=very poor; 2=poor; 3=fair; 4=good; 5=very good. The overall percentage score was computed as a sum of items 1 to 14 as expressed as a percentage of the maximum possible score: Overall Percentage Score = Sum [item 1... item 14]-14)/(70-14 ) *100%. Q-LES-Q overall percentage score can range from 0 to 100, with higher values indicating higher quality of life.
Time Frame: Baseline, Weeks 2, 4, 6, 8, based on last observation carried forward (LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
units on a scale
  Baseline | 52.4 (14.9) | 52.2 (13.5) | 52.0 (14.8)
  Week 2- Change from baseline | 3.1 (10.6) | 2.1 (13.2) | 1.5 (12.1)
  Week 4- Change from baseline | 4.7 (12.4) | 5.4 (12.7) | 4.6 (12.8)
  Week 6- Change from baseline | 5.8 (13.7) | 6.7 (13.4) | 5.0 (13.6)
  Week 8- Change from baseline | 7.0 (14.8) | 6.8 (13.2) | 5.8 (14.6)

9. Secondary Outcome: Change From Baseline Insomnia Severity Index (ISI) Total Score
Description: The ISI was completed by the subject and is an assessment of the severity of insomnia. The administered extended ISI questionnaire consists of 5 items (containing 7 questions, as item 1 contains 3 questions) comprising the original ISI questionnaire, plus 6 quality of life related items (sleep quality, restedness/refreshness upon arising, daytime fatigue, attention/concentration, relationships and mood disturbances), and 2 items assessing duration and frequency of sleep problems. All items, except for the insomnia duration and frequency questions, are measured on a Likert-type 5-point scale (0-4). ISI total score can range from 0 to 28, with higher scores indicating more severe insomnia.
Time Frame: Baseline, Weeks 2, 4, 6, 8, based on lst observation carried forward (LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
units on a scale
  Baseline | 14.6 (5.3) | 14.3 (5.3) | 14.1 (6.0)
  Week 2- Change from baseline | -2.4 (4.4) | -1.5 (5.0) | -2.7 (5.3)
  Week 4- Change from baseline | -3.6 (4.8) | -3.1 (5.4) | -3.4 (5.3)
  Week 6- Change from baseline | -4.0 (5.6) | -3.6 (5.5) | -3.6 (5.6)
  Week 8- Change from baseline | -4.3 (5.6) | -3.5 (6.2) | -4.1 (5.8)

10. Secondary Outcome: Change From Baseline Sheehan Disability Scale (SDS)
Description: The SDS was completed by the subject and captured the subject's level of disability. The subject rated the extent to which his or her work, social life or leisure activities, and home life or family responsibilities were impaired by his or her symptoms on a 10-point visual analog scale. SDS total score can range from 0 to 30, with higher scores indicating higher functional impairment.
Time Frame: Baseline, Weeks 2, 4, 6, 8, based on last observation carried forward (LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
units on a scale
  Baseline | 15.3 (6.7) | 14.0 (6.4) | 14.8 (6.4)
  Week 2- Change from baseline | -2.5 (5.5) | -0.9 (6.3) | -2.7 (5.3)
  Week 4- Change from baseline | -3.6 (6.1) | -2.5 (6.3) | -3.5 (6.1)
  Week 6- Change from baseline | -4.2 (6.5) | -3.4 (6.3) | -4.1 (6.2)
  Week 8- Change from baseline | -5.1 (6.6) | -4.1 (6.5) | -4.4 (6.2)

11. Secondary Outcome: Change From Baseline Epworth Sleepiness Scale (ESS)
Description: ESS was completed by the subject and assessed daytime sedation based on 8 items, each presenting a situation for which the subject needed to evaluate how likely he/she is to doze off or fall asleep in contrast to feeling just tired. Each item was evaluated on the following scale: 0 = would never doze; 1 = slight chance of dozing; 2 = moderate chance of dozing; 3 = high chance of dozing. ESS total score can range from 0 to 24, with higher scores indicating higher levels of daytime sleepiness.
Time Frame: Baseline, Weeks 2, 4, 6, 8, based on last observation carried forward (LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Number analyzed (Participants) | 149 | 146 | 145
units on a scale
  Baseline | 7.4 (4.5) | 8.4 (4.5) | 8.5 (4.8)
  Week 2- Change from baseline | -0.1 (4.0) | -0.5 (3.8) | -0.4 (3.6)
  Week 4- Change from baseline | -0.2 (4.6) | -1.0 (4.1) | -0.7 (4.5)
  Week 6- Change from baseline | -0.6 (4.0) | -1.3 (4.0) | -0.9 (4.5)
  Week 8- Change from baseline | -0.8 (4.0) | -1.4 (4.2) | -1.3 (4.5)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebo Arm | Eszopiclone Low Dose Arm | Eszopiclone High Dose Arm
Serious Adverse Events (participants affected / at risk) | 0/149 | 3/146 | 0/145
Other Adverse Events (participants affected / at risk) | 104/149 | 111/146 | 116/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=149) | Eszopiclone Low Dose Arm (N=146) | Eszopiclone High Dose Arm (N=145)
Amniotic Cavity Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Self Injurious Behavior (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=149) | Eszopiclone Low Dose Arm (N=146) | Eszopiclone High Dose Arm (N=145)
Nausea (Gastrointestinal disorders) | 14 (19) | 7 (8) | 18 (21)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 5 (5) | 13 (16)
Dry Mouth (Gastrointestinal disorders) | 6 (7) | 8 (8) | 12 (12)
Abdominal Pain Upper (Gastrointestinal disorders) | 10 (11) | 9 (12) | 14 (20)
Fatigue (General disorders) | 12 (14) | 12 (12) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 12 (12) | 4 (4)
Nasaopharyngitis (Infections and infestations) | 5 (6) | 6 (6) | 8 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (11) | 4 (5)
Headache (Nervous system disorders) | 27 (47) | 26 (44) | 24 (41)
Dysgeusia (Nervous system disorders) | 3 (3) | 10 (16) | 35 (37)
Dizziness (Nervous system disorders) | 6 (7) | 11 (15) | 16 (20)
Somnolence (Nervous system disorders) | 7 (7) | 8 (8) | 10 (11)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish